CLINICAL TRIAL: NCT04213586
Title: Effects of Whey Protein and Collagen Supplementation on Muscle Mass and Function During Training in Young Adults
Brief Title: Effects of Whey Protein and Collagen Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Collaborators: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Andreo Fernando Aguiar, Principal Investigator, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 3.058.958
Record Dates: First submitted 2019-12-11; First posted 2019-12-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Exercise; Nutrition Therapy; Resistance Training; Muscle Strength; Hypertrophy
Keywords: Protein supplementation; Amino acids; Resistance exercise; Muscle strength; Muscle hypertrophy
MeSH Terms: conditions — Motor Activity; Hypertrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey Protein (Experimental): Each participant will be supplemented with whey protein (7 d/wk) during 10 weeks.
  Interventions: Dietary Supplement: Whey protein supplementation
- Leucine-matched collagen (Experimental): Each participant will be supplemented with collagen (7 d/wk) during 10 weeks.
  Interventions: Dietary Supplement: Collagen supplementation

INTERVENTIONS:
Dietary Supplement: Whey protein supplementation — 35 g of whey protein (7 d/wk) during a 10-wk resistance training program (3 d/wk; 3 sets of 8-12 repetitions with an interval of 1-2 minutes between sets and exercises) involving the leg press, leg extension, and arm flexion exercises. The load will be adjusted weekly.
  Arms: Whey Protein
Dietary Supplement: Collagen supplementation — 35 g of collagen (7 d/wk) + 2 g of leucine during a 10-wk resistance training program (3 d/wk; 3 sets of 8-12 repetitions with an interval of 1-2 minutes between sets and exercises) involving the leg press, leg extension, and arm flexion exercises. The load will be adjusted weekly.
  Arms: Leucine-matched collagen

SUMMARY:
The present project aims to investigate the effects of high-quality protein (whey protein) vs. low-quality protein (collagen) on muscle mass and function (e.g., strength and power) during a 10-wk resistance training program in young adults. It will be tested the hypothesis that leucine-matched collagen should promote similar gains on muscle function and mass compared to whey protein supplementation.

DETAILED DESCRIPTION:
The purpose of this study will be to investigate the effects of whey protein vs. leucine-matched collagen supplementation on muscle mass and function after a 10-wk resistance training program. Initially, all participants will be submitted for a 2-wk familiarization period, and then randomized into two groups (N = 11 / group): whey protein group and leucine-matched collagen group. The following variables will be assessed from pre-to post-training: anthropometric, muscle thickness from vastus lateralis and biceps brachii muscles using ultrasound, training load, mean power and peak torque for unilateral arm flexion exercise using a isokinetic dynamometer, countermovement vertical jump, nutritional intake, and testosterone-to-cortisol ratio . Shapiro-Wilk and Levine tests will be used to test the normality and homogeneity of the measurements, respectively. Two-way ANOVA (group x time) tests for repeated measures will be performed to assess changes over time and between groups for all dependent variables. Violation of sphericity will adjust using Greenhouse- Geyser correction. The Bonferroni post-hoc test will detect specific differences between groups. When appropriate, the percentage of change (∆%) will be reported according to the following equation: ∆% = [(pre-average post average) / pre-average mean] × 100. Values will be express as mean ± standard deviation. O significance level α will be 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-35 years
* To be eutrophic (not overweight or obese)

Exclusion Criteria:

* To present a history of musculoskeletal disorders
* Be attending a systematized weight training program for at least six months
* To make use of medicines that could affect muscle function.
* To have used ergogenic supplements and anabolic steroids for at least six months before study
* To have restrictions for exercises practice considering Physical Activity Readiness Questionnaire (PAR-Q) responses.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Change in biceps brachii thickness | Baseline and after 10 weeks
  Measured by ultrasonography pre- and post-training
Change in muscle strength by training load | Baseline, 5 and 10 weeks
  Training load for leg press, knee extension, and arm flexion exercises
Change in vertical jump | Baseline and after 10 weeks
  Countermovement vertical jump performance will be assessed using the Smart Jump instrument
Change in mean power | Baseline and after 10 weeks
  Mean power using a isokinetic dynamometer (BIODEX)
Change in peak torque | Baseline and after 10 weeks
  Peak torque using a isokinetic dynamometer (BIODEX)
Change in vastus lateralis thickness | Baseline and after 10 weeks
  Measured by ultrasonography pre- and post-training

SECONDARY OUTCOMES:
Change in testosterone-to-cortisol ratio | Baseline and after 10 weeks
  Blood samples will be collected for analyse of the testosterone-to-cortisol ratio
Dietary intake | Baseline, 2, 5, 10 weeks
  Dietary intake to be assessed using 3-day diet recalls.

CONTACTS AND LOCATIONS:
Overall Officials: Andreo Aguiar, Principal Investigator — Universidade Norte do Paraná
Locations (1):
- Universidade Norte do Paraná, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No